CLINICAL TRIAL: NCT03189940
Title: Effect of Lifestyle Modification Using Smartphone Application on Weight Reduction and Obstructive Sleep Apnea
Brief Title: Lifestyle Modification Using an App in OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Whun Kim, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-1504-296-302
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Obstructive Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App user group (Active Comparator)
  Interventions: Behavioral: Life style modification by using and app with a wrist-worn activity tracker
- Control group (Sham Comparator): Control participants, the physicians could assess the lifestyle and recommend further lifestyle modification only on the basis of the participants' recalls
  Interventions: Behavioral: Conventional Life style modification

INTERVENTIONS:
Behavioral: Life style modification by using and app with a wrist-worn activity tracker — The mobile app was designed to collect daily lifestyle data by wearing a wrist activity tracker and reporting dietary intake. At the visit after 2 weeks of use, a summary of the lifestyle was displayed on the hospital EMR and reviewed by both physicians and app users. Further lifestyle modification was encouraged on the basis of the electronically collected data.
  Arms: App user group
Behavioral: Conventional Life style modification — Physician's usual consultation for life style modification at 0 week, and 2 weeks of enrollment
  Arms: Control group

SUMMARY:
This study aimed to investigate the effects of a mobile phone app linked to hospital electronic medical record (EMR) system on weight reduction and obstructive sleep apnea (OSA). Adults aged > 20 years with witnessed snoring or sleep apnea from a sleep clinic of a tertiary center were prospectively enrolled, and the participats were randomized into app user and control groups. The mobile app was designed to collect daily lifestyle data by wearing a wrist activity tracker and reporting dietary intake. At the visit after 2 weeks of use, a summary of the lifestyle was displayed on the hospital EMR and reviewed by both physicians and app users. Further lifestyle modification was encouraged on the basis of the electronically collected data. In the control group, the lifestyle modification performed as the usual practice. All participants underwent Watch PAT and body mass index (BMI) measurement twice: on enrollment; and after 4-weeks follow up. Changes of BMI, and parameters of sleep related breathing were analyzed.

ELIGIBILITY:
Inclusion Criteria:

ᆞ patients must agree to participate in our clinical study ᆞ patients without severe cardiopulmonary disease ᆞ patients must be with BMI > 23 Kg/m2

Exclusion Criteria:

ᆞ patients who did not agree ᆞ patients with severe cardiopulmonary disease ᆞpatients who are under treatment using a continuous positive airway pressure device or a mandibular advancement device ᆞ patients who were pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-11-18 (Actual)

PRIMARY OUTCOMES:
changes in body weight | base line and after 4weeks of life style modiciation
  body weight measurement and calculate into body mass index (BMI)

SECONDARY OUTCOMES:
apnea hypopnea index (AHI) | base line and after 4weeks of life style modiciation
  number of apnea and or hypopnea event per hour during sleep
respiratory distress index (RDI) | base line and after 4weeks of life style modiciation
  AHI + number of respiratory effor related arousal (RERA) per hour during sleep
oxygen desaturation index (ODI) | base line and after 4weeks of life style modiciation
  number of desaturation event (peripheral oxygen satuation less than 90%) per hour during sleep
sleep time proportion with snoring loudness > 45dB | base line and after 4weeks of life style modiciation
  total duration of the snoring loudness >45 dB devided by the total sleep time (%)
lowest oxygen saturation | base line and after 4weeks of life style modiciation
  the degree of the lowest oxygen saturation measured during sleep

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Whun Kim, MD, PhD, Study Director — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No
the individual data is confidential according to the hospital's policy